CLINICAL TRIAL: NCT05309122
Title: A Retrospective Cohort Study on the Effectiveness of Various Screening Strategies for Uterine Cervical Cancer
Brief Title: Cervical Cancer Screening Strategies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EVUCC
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia; Human Papillomavirus Infection; Cervical Cytology; Cancer Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Cervical exfoliated cells collected by pap smear or by Thinprep cytology testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to investigate retrospectively the results of cervical cytology and high-risk human papillomavirus in the past 20 years recorded in Peking Union Medical College Hospital. The histological findings after cervical cancer screening were reviewed. The diagnostic values of different screening strategies were compared based on the results of cervical histology. The primary endpoint is the diagnosis of grade 2 cervical intraepithelial neoplasia (CIN2) or more severe lesions (CIN2+). The secondary endpoints include following objectives: (1) the invasive procedures needed according to the screening results; (2) the diagnosis of vaginal and/or vulval intraepithelial neoplasia; (3) the persistence and recurrence of human papillomavirus infection; and (4) the cost-effectiveness of screening strategies for CIN2+.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* With definite cervical histology after cervical cancer screening, ore with at least one screening test after first testing

Exclusion Criteria:

- Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who accepted cervical cancer screening in the study center
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-03-19 (Actual); Primary Completion 2024-03-19 (Estimated); Study Completion 2025-03-19 (Estimated)

PRIMARY OUTCOMES:
CIN2+ | One year
  CIN2+ detected by various screening methods

SECONDARY OUTCOMES:
Invasive procedures | One year
  Invasive procedures needed according to the screening results
Vaginal intraepithelial neoplasia (VaIN) | One year
  VaIN detected by various screening methods
Vulval intraepithelial neoplasia (VIN) | One year
  VIN detected by various screening methods

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China